CLINICAL TRIAL: NCT02960009
Title: Motor Excitability Study of High Definition Transcranial Direct Current Stimulation (HD-tDCS) in Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2015.691-T
Record Dates: First submitted 2016-09-14; First posted 2016-11-09 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anode HD-tDCS (Experimental): The center anode is fixed on the ipsilesional primary motor cortex and the 4 surrounding cathode electrodes will be placed about 6 cm to the center.
  Interventions: Device: HD-tDCS
- Cathode HD-tDCS (Experimental): The center cathode is fixed on the contralesional primary motor cortex and the 4 surrounding anode electrodes will be placed about 6 cm to the center.
  Interventions: Device: HD-tDCS
- Sham HD-tDCS (Placebo Comparator): The center anode is fixed on the ipsilesional primary motor cortex and the 4 surrounding cathode electrodes will be placed about 6 cm to the center.
  Interventions: Device: HD-tDCS

INTERVENTIONS:
Device: HD-tDCS — Different stimulation protocols will be applied to the primary motor cortex of stroke patients. After 20-minute stimulation, EMG-driven robot hand training will be conducted.

SUMMARY:
High definition tDCS will be conducted to both stroke and healthy subjects on primary motor cortex area to explore the motor excitability changes before and after stimulation. In next stage, a randomized control trial with 20-session training will be conducted to evaluate the effectiveness of transient modulation of cortical excitability through multisite HD-tDCS with EMG driven robot hand training, a sham stimulation with EMG-driven robot hand training will be applied as control group.

ELIGIBILITY:
Inclusion Criteria:

1. Sufficient cognition to follow simple instructions, as well as understand the content and purpose of the experiment;
2. Have moderate to severe motor disability at the paretic upper limb (assessed by Fugl-Meter Assessment (FMA), and Action Research Arm Test (ARAT));
3. Hemiparesis resulting from a single unilateral lesion of the brain with onset at least 6 months before data collection

Exclusion Criteria:

1. Severe hand spasticity, open hand wound or hand deformity;
2. Visual field deficits;
3. Aphasia, neglect, and apraxia;
4. History of alcohol, drug abuse or epilepsy;
5. Bilateral infracts;
6. Uncontrolled medical problems;
7. Serious cognitive deficits [Mini-Mental State Examination (MMSE) < 21];
8. Major depression
9. Metal implants inside body
10. MRI, TMS and tDCS contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography (EEG) and Electromyography (EMG) | Before intervention, During intervention, After intervention, 6-month after intervention
  It is used to investigate the changes in corticomuscular coherence for studying connectivity between the brainwave using EEG and the affected hand muscles using EMG. In addition, EMG will be used to detect muscle activation change and muscle co-contraction pattern alteration.
Action Research Arm Test (ARAT) | Before intervention, After intervention, 6-month after intervention
  The ARAT is a 19-item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement) to assess upper limb functioning
Fugl-Meyer Assessment Upper Extremity (FMA-UE) | Before intervention, After intervention, 6-month after intervention
  It is used to evaluate and measure upper-limb recovery in post-stroke hemiplegic patients, and items are scored on a 3-point ordinal scale

SECONDARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | Before intervention, After intervention, 6-month after intervention
  It is used to identify neural correlates of stimulation-induced behavioral gains for investigating tDCS-induced changes in brain activations
Transcranial Magnetic Stimulation (TMS) | Before intervention
  It is used to measure the changes in interhemispheric imbalance and corticospinal excitability

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kai-yu Tong, PhD, Principal Investigator — Department of Biomedical Engineering, CUHK
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No